CLINICAL TRIAL: NCT03231475
Title: Phase I, Open-label Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of SPH1188-11 Tablets for the Treatment of Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC).
Brief Title: Phase I Study of SPH1188-11 in NSCLC
Acronym: SPH1188-11
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Board decision
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH1188-11-101
Record Dates: First submitted 2017-06-06; First posted 2017-07-27 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: NSCLC Stage IIIB; NSCLC Stage IV
Keywords: NSCLC; EGFR-TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPH1188-11 (Experimental): SPH1188-11 dose escalation, 50mg/100mg/200mg/300mg/450mg/600mg
  Interventions: Drug: SPH1188-11

INTERVENTIONS:
Drug: SPH1188-11 — qd.po
  Other Names: SPH1188

SUMMARY:
This study will treat patients with advanced NSCLC who have already received at least one course of specific anti-cancer treatment but the tumour has started to re-grow following that treatment. This is the first time this drug has ever been tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment, it will measure the levels of drug in the body, it will also measure the anti-cancer activity. By using these pieces of information together the best dose of this drug to use in further clinical trials will be selected.

DETAILED DESCRIPTION:
Phase I dose escalation study

ELIGIBILITY:
Inclusion Criteria:

1. 18-70years old, male or female.
2. Histological or cytological confirmation diagnosis of Non Small Cell Lung Cancer(NSCLC),Stage IIIBorIV, previous treatment with 1st EGFR-TKI, and/or previous chemotherapy. Regardless of EGFR mutation status.
3. At least one measurable disease according to RECIST 1.1.
4. Life expectancy of at least 3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
6. Females should be using adequate contraceptive measures from the time of screening until 3 months after discontinuing study treatment, should not be breast feeding and must have a negative pregnancy test 7days prior to start of dosing. Males should be willing to use barrier contraception during the trial and 3 months after discontinuing study treatment.
7. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.

Exclusion Criteria:

1. Treatment with an EGFR-TKI(eg, erlotinib, gefitinib, icotinib) within 7 days or approximately 5x half-life of study entry.
2. Previous treatment with 2nd EGFR-TKI or 3rd EGFR-TKI(eg, afatinib, osimertinib).
3. Any cytotoxic chemotherapy or anticancer drugs within 4 weeks of the first dose of study treatment.
4. Major surgery(excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
5. Radiotherapy within 4 weeks of the first dose of study treatment.
6. Patients currently receiving(or unable to stop use at least 1 week prior to receiving the first dose) medications or herbal supplements known to be potent inhibitors of CYP3A4/CYP2D6, and/or potent inducers of CYP3A4/CYP2D6.
7. Laboratory values within 7 days of the first dose of study treatment:

   * Absolute neutrophil count<1.5×10^9/L
   * Platelet count <100×10^9/L
   * Haemoglobin<90 g/L
   * Alanine aminotransferase>2.5 times the upper limit of normal(ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
   * Aspartate aminotransferase>2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
   * Total bilirubin>1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome(unconjugated hyperbilirubinaemia) or liver metastases.
   * Creatinine>1.5 times ULN concurrent with creatinine clearance <50ml/min(measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is>1.5 times ULN.
8. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events(CTCAE) grade 1 at the time of starting study treatment (except alopecia and prior platinum-therapy related neuropathy)
9. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
10. Any evidence of severe or uncontrolled systemic diseases, including active bleeding, active infection including hepatitis B(HBsAg+ and HBV-DNA+), hepatitis C and human immunodeficiency virus(HIV).
11. Cardiac criteria: QTc>480msec. LVEF<50%. Any clinically important abnormalities in rhythm, any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family in first degree relatives or any concomitant medication known to prolong the QT interval.
12. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
13. Idiopathic pulmonary fibrosis.
14. Chronic gastrointestinal diseases, characterized by diarrhea.
15. Inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of SPH1188-11.
16. History of Keratitis, ulcerative keratitis, severe xerophthalmia.
17. Previous or concomitant malignancies at other sites, except effectively treated nonmelanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 5 years and is considered to be cured.
18. History of neurological or mental disorders, including epilepsy or dementia.
19. Allergy to the test drug or any excipient of the product.
20. Participate in other drug clinical trials within 4 weeks of the first dose of study treatment.
21. Receiving any other anti-tumor therapy.
22. Women who are breast feeding or pregnant.
23. Judgment by the investigator that the patient should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
DLT and MTD of SPH1188-11 | 28 days
  Incidence and intensity of Adverse Events according to Common Toxicity Criteria (CTC version 4.03) associated with increasing doses of SPH1188-11, to find DLT and MTD

SECONDARY OUTCOMES:
Tmax of SPH1188-11 | 28 days
  Evaluate the Tmax of SPH1188-11
ORR of SPH1188-11 | 52 weeks
  Objective response rate(ORR) according to RECIST 1.1, ORR=CR+PR
PFS of SPH1188-11 | 52 weeks
  Progress free survival(PFS)
DCR of SPH1188-11 | 52 weeks
  Disease control rate(DCR), DCR=CR+PR+SD
Cmax of SPH1188-11 | 28 days
  Evaluate the Cmax of SPH1188-11
AUC of SPH1188-11 | 28 days
  Evaluate the AUC of SPH1188-11
T1/2 of SPH1188-11 | 28 days
  Evaluate the T1/2 of SPH1188-11

CONTACTS AND LOCATIONS:
Overall Officials: JunNing Cao, Master, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No